CLINICAL TRIAL: NCT03638154
Title: Clinical Regenerative Potential of Cultured Gingival Fibroblast- Mesenchymal Stem Cells in Treatment of Periodontal Intrabony Defects (Randomized Clinical and Biochemical Trial)
Brief Title: Regenerative Potential of Cultured Gingival Fibroblast- Mesenchymal Stem Cells in Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mahetab mohamed abdel el wahab, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER 16-P1
Record Dates: First submitted 2018-06-22; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Periodontal Intrabony Defect

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupI (Placebo Comparator): safety with received beta-tricalcium phosphate (β TCP) bone substitute only. (Bioresorb, Sybron, implant solutions GmbH Bremen, Germany)
  Interventions: Procedure: β TCP bone substitute only
- GroupII (Active Comparator): safety with surgical augmentation of GF+GMSCs carried on β TCP in intrabony periodontal defect and covered by collagen membrane and received a mixture of gingival fibroblast(GF) and gingival mesenchymal stem cells(GMSCs) carried on a vehicle of β TCP covered by a resorbable collagen membrane.
  (Cytoplast, RTM Collagen Cytoplast, Barrier Membranes, Osteogenics Biomedical, New Jersey, USA).
  Interventions: Procedure: GF+GMSCs carried on β TCP

INTERVENTIONS:
Procedure: GF+GMSCs carried on β TCP — surgical augmentation of GF+GMSCs carried on β TCP in intrabony periodontal defect and covered by collagen membrane(Bioresorb, Sybron, implant solutions GmbH Bremen, Germany) Cytoplast, RTM Collagen Cytoplast, Barrier Membranes, Osteogenics Biomedical, New Gersey, USA).
  Ibuprofen
  Arms: GroupII
Procedure: β TCP bone substitute only — surgical augmentation by β TCP in intrabony periodontal defect(Bioresorb, Sybron, implant solutions GmbH Bremen, Germany) Ibuprofen
  Arms: GroupI

SUMMARY:
clinical trial was conducted to evaluate regenerative potentials of cultured gingival fibroblasts and GMSCs carried in beta tri calcium phosphate scaffold into intrabony periodontal defects in human by clinical and radiographic parameters

DETAILED DESCRIPTION:
In the present study, twenty posterior two or three osseous intrabony periodontal defects were involved . They were grouped in to two groups. Group I included ten intrabony posterior defect received beta tri calcium phosphate (β TCP) bone substitute. Group II included ten posterior intrabony periodontal defect and they received a mixture of gingival fibroblast(GF) and gingival mesenchymal stem cells(GMSCs) carried on a vehicle of β TCP covered by a resorbable collagen membrane. CBCT was used preoperatively and after 6 months for hard tissue evaluation. PDGF and BMP were measured in GCF at days 1,3,7,14.

ELIGIBILITY:
Inclusion Criteria:

* Presence of interproximal osseous defects estimated from radiographic evaluation (Cone Beam CT) and transgingival bone sounding ≥3mm of two or three osseous walls.

  * Probing Depth ≥5mm after initial therapy.
  * Attachment loss ≥4mm.
* full mouth plaque score and bleeding on probing score ≤ 20% after phase I therapy.

  * non vital teeth only involved.
  * no furcation involvement of the teeth presenting the intraosseous defects.
  * Thick gingival biotype more than 1 mm with enough width of attached gingiva.
* Accepts Healthy Volunteers

Exclusion Criteria:

* Patients with systemic disease or compromised immune illness using Cornell medical index
* Smoker's patients.
* Pregnant and lactating females.
* Uncooperative patients (low compliance, bad oral hygiene).
* Decision impaired individuals (prisoners, handicapped and mentally retarded patients).

Ages: 32 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
bone gain in periodontal defects(by mm) | 6 months
  20 patients were involved as assessed by cone beam ct at baseline (pre) and 6 months later(post). the fusion of pre and post operative cone beam ct scan of the intrabony periodontal defect to measure bone gain by mm. so that, the regenerative potentials of cultured gingival into ten intrabony defect fibroblasts and GMSCs carried by tri calcium phosphate , the bone gain was measured by radiographic fusion of pre and post image of intrabony periodontal defects in human.

SECONDARY OUTCOMES:
the regenerative power of the defect was evaluated by growth factor concentration in GCF. | day 1,3,7,14 after surgery
  4 GCF samples were collected from each patient at day 1,3,7,14 after periodontal surgery then a Biochemical analysis of BMP-2 and PDGF-bb (by mg /dl) concentrations in GCF by using ELIZA kite which reflect the healing power at the initial periods of healing in different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gamal, professor, Study Director — Professor of Oral Medicine, Periodontology and Oral Diagnosis, Faculty of Dentistry, Ain Shams University

DOCUMENTS (1):
  • Study Protocol (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT03638154/Prot_000.pdf